CLINICAL TRIAL: NCT07110077
Title: Implementing a Young First Aiders (YoFA) Training Program Amongst Early Secondary School Children on Injury and Trauma First Aid in Fako Division.
Brief Title: Pre and Post-Implementation of Injury/Trauma First Aid Training Among Early Secondary School Students in Fako, Cameroon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Buea (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Tabe Orock-Benem Vanessa, PhD fellow/Principal Investigator, University of Buea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 029/CRERSH/SW/C/11/2024; D43TW012186 (NIH)
Record Dates: First submitted 2025-07-21; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Trauma/Injury Problem
Keywords: Trauma/injury First aid; secondary school children; Young First Aiders (YoFA)
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The intervention group will be trained on fundamental aspects of First Aid with a special focus on identifying and stopping life-threatening bleeds. The students will be trained in 4 groups of 20 students. Training will last 5 hours over 2 days, spread over 2 weeks. That is, once a week on the days during which they have a "half-day" of classes. Afterward, these will be followed up on a biweekly basis for 3 months before a final evaluation is made. We would also do an adapted system usability scale to see how usable the skills taught to the students were and the ease of use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training of Young First Aiders in secondary schools (Experimental): There is just one arm which has already been described. The control group will just be observed with no intervention given.
  Interventions: Other: Young First Aiders Traing of Early Secondry School children

INTERVENTIONS:
Other: Young First Aiders Traing of Early Secondry School children — Training Young First Aiders in Early Secondary School Children with a pre-, immediate post- and final post-tests to determine knowledge change.

SUMMARY:
To save lives, alleviate pain, and prevent injuries from worsening before medical assistance can be summoned, first aid is essential. These fundamental skills are accessible to everyone, including young people. Worldwide, first aid training has consistently improved outcomes and reduced injury-related complications. Although first aid training for adults is widely available, it is equally important to equip young people in schools with these skills so they can defend themselves and support their communities.

'Young First Aiders' (YoFA) is a youth-specific first aid program that is the subject of this study, to be conducted in the Fako Division, Cameroon. Its primary goals are to:

* Determine how stakeholders view the YoFA program.
* Assess whether YoFA enhances the knowledge, attitudes, and practices (KAP) of first aid among secondary school pupils.
* Determine the difficulties in providing this age group with first aid training.
* Assess the program's overall usefulness and efficacy.

The investigator will use a mixed-methods approach for the study in the Tiko and Buea health districts. It entails gathering extensive data via:

Focused group discussions, surveys, interviews, and scenario observations. To enable a direct comparison of results, one district will act as the intervention group and receive the YoFA training, while the other will act as the control group. To obtain a variety of viewpoints on the program, researchers will interview a large number of participants, including parents, educators, students, and administrators. Participants will complete customized surveys, which will be analyzed using Dedoose and R software to examine qualitative data from observations and interviews.

Expectations of this study include: Identifying barriers to making first aid instruction for children 10 to 14 years old successful, creating solutions to deal with these issues that have been identified. Moreover, to see if YoFA participants' first aid skills have improved, including their capacity to stay safe in an emergency, call for help, and offer prompt assistance (such as halting potentially fatal bleeding).

All this, to increase youth access to first aid training, which will help them develop a culture of readiness and self-assurance in managing crises as they get older; hence building a growing first aid culture to handle prehospital care.

DETAILED DESCRIPTION:
PROBLEM STATEMENT Due to its limited inclusion in medical and educational curricula, first aid (FA) knowledge and practice are severely lacking, particularly in sub-Saharan Africa and Cameroon. According to WHO data, the majority of schools do not have operational dispensaries, and there is a serious shortage of medical personnel. Improvements in school health facilities have not kept up with the rise in student enrollment, and there are insufficient systems in place for referring students to medical facilities. It is essential to increase FA awareness among teachers and students, who are frequently the first to respond to incidents. FA skills can be improved and formal training may be encouraged in the future by implementing programs like YoFA with continuous refresher courses.

RESEARCH QUESTIONS

1. What community perceptions exist about children learning and/or using FA skills within the school setting or thereabouts?
2. What is the level of Knowledge, the attitudes and practices (KAP) of early secondary school children (SSC) on injury/trauma FA?
3. How efficacious and usable is an injury/trauma Young First Aiders' (YoFA) training program to early SSC and the community?
4. What are the perceived barriers/challenges and benefits of the YoFA program in schools and the community?

RESEARCH OBJECTIVES General Objective

1. To gain insights into the perceptions and barriers surrounding a Young First Aiders' (YoFA) training program on trauma/injury first aid in both the school setting and the community in the Fako Division.
2. To assess and measurably improve KAP of SSC on trauma/injury FA using the YoFA training program in Fako Division.

Specific Objectives

1. To understand the perspectives of stakeholders (school teachers, administrators, parents, community leaders and students) on a school-based FA training (YoFA) program among SSC.

   Hypothesis 1: The perspectives of stakeholders like school administrators, teachers, parents, community leaders, and school children needs to be understood to design a comprehensive YoFA program
2. To assess school children's Knowledge, Attitudes (willingness to) and Practices (self-efficacy) (KAP) on trauma/injury FA via the built YoFA training to stop LTBs.

   Hypothesis 2: School children have limited knowledge, self-efficacy and practices regarding trauma/injury FA
3. To evaluate the effectiveness and usability of the YoFA training program for SSC to respond to LTBs safely and promptly in their environs.

   Hypothesis 3: The YoFA training Program is effective in improving the KAP of SSC and it is usable within the school and community setting.
4. To determine the barriers associated with implementing the YoFA program among early SSC in the Fako Division.

Hypothesis 4: There exist some barrier/challenges in implementing a YoFA training program in secondary schools.

METHODOLOGY

STUDY AREA:

The Southwest region is one of the two (2) English speaking regions of the 10 regions in Cameroon. These regions have been in some socio-political crises for seven (7) years now and there have been an increase in road traffic crashes and injuries for which prehospital care would have helped. But the absence of it and worsening of road conditions calls for more action geared towards prehospital care than not. The investigators saw this need and decided to build a first aid culture starting from the young. Fako division is one of the most accessible divisions due to the conflict in the Southwest with four (4) health districts; Buea, Limbe, Tiko and Muyuka. The Buea and Tiko Health Districts will be selected based on the district with the highest number of trauma cases recorded in the DHIS2 and the security situation within the region.

The highest number of trauma from 2020 to 2023 were 488,494,375, and 1281 for Buea Limbe, Muyuka and Tiko respectively. After Tiko, although Limbe is the next district with the next highest number of trauma and injury cases after Tiko, the investigators took Buea to avoid the confounding effects of the Lay First-responders (LFR) program taking place in Limbe

Study population:

The study population includes various stakeholders for the qualitative part, such as teachers, parents, school administrators and students in Buea and Tiko. The cross-sectional survey and intervention will focus on early secondary school students (Forms 1-3) aged 10-14, who are transitioning from primary school. The evaluation will involve students to assess the program's impact, challenges, and the need for refresher courses STUDY DESIGN A mixed-methods exploratory sequential approach, incorporating both quantitative surveys and qualitative interviews.

Qualitative part:

The investigator and trained research assistants will do focused group discussions (FGDs) with parents, teachers, school administrators and students in groups of 5 to 12. From those, 2 other participants per group will be interviewed in-depth (IDIs). All these FGDs and IDIs will take place within the school campuses.

Quantitative Part:

The quantitative aspect will take part within the school campuses and involve administering questionnaires to students to assess their knowledge, attitudes (confidence), and practices (utilization/usability) of FA trauma/injury skills before and after their training. This will focus mostly on staying safe, calling for help and stopping a life-threatening bleed. The intervention will include training the intervention group in reasonable clusters of 15 to 20 students per group for 2.5 hours per day for 2 days in 2 weeks. Following this, a biweekly follow up will be performed with physical reminders of the group of students. The control will have no intervention.

The students will be trained within the school premises on Wednesdays, given that they have school half days then. The student participants will be followed up for 3 months after the main training sessions.

Sample Size Calculation Calculated at 134 participants for both the intervention and control groups (67) per group.

All assumptions considered are seen in the main protocol.

ELIGIBILITY:
Inclusion Criteria:

* For the Quantitative part
* Form one (1) to three (3) students (ages 10 to 14 years) in five (5) state secondary schools (SSS) in Tiko and Buea health districts who are willing to participate in the study.
* Students officially enrolled in the school for the academic year
* Those students whose parents consent for their children to be part of the study.

For the Qualitative part

* Stakeholders within the educational care system - students, school teachers and school administrators (e.g., (Principals) community stakeholders (parents) who consent to be part of the study.
* Students whose parents give parental consent for their children to participate in the study.

Exclusion Criteria:

* Any child who is not in forms 1 to 3 (10 to 14 years old) in the selected schools
* Any student who misses any of the training sessions
* Any student who willingly backs out of the study.
* Any child whose parents do not give parental consent for them to be part of the study

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Change in Knowledge on Injury and trauma first aid | Baseline, 2 weeks and 3months
  To help us determine the knowledge change before the training, immediately ater and 3 months after the training. A score was assigned to the pre- and post-tests on 24 points for the 24 knowledge, attitude and practice questions and converted to percentage. the change in knowledge from pre to post test is measured to see whether there was a change in first aid knowledge
Change in knowledge | Baseline, two weeks, and 3 months
  Determine the knowledge change before, immediately after and 3 months after the training. A score was assigned to the pre- and post-tests on 24 points for the 24 knowledge, attitude and practice questions and converted to percentage. the change in knowledge from pre to post test is measured to see whether there was a change in first aid knowledge

SECONDARY OUTCOMES:
Number of Participants who used/ thought the the skills taught after the training were usable. | End of the 3-month post-test.
  A 10-point adapted System Usability Scale in Likert format is used to collect this information.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Chichom Mefire, Professor of Surgery, Study Chair — University of Buea; Ariane Christy Sabrinah, MD, Study Director — University of California
Locations (1):
- University of Buea, Buea, Southwest Region, Cameroon

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie result
Supporting Information: Study Protocol, ICF
Time Frame: January 2025 to January 2026
Access Criteria: Leaders of the scientific review committee for the journal that will be responsible for publishing results of the study. They will be able to access consent forms and questionnaires used for data collection upon sending a request to the PI for this information using the link that will be provided.
URL: https://drive.google.com/drive/folders/1oaz8ewLKW--cX5Nm7Y0I_j0jPhJzwzVS?usp=sharing

REFERENCES:
- [Background] Joseph N, Kumar G, Babu Y, Nelliyanil M, Bhaskaran U. Knowledge of first aid skills among students of a medical college in mangalore city of South India. Ann Med Health Sci Res. 2014 Mar;4(2):162-6. doi: 10.4103/2141-9248.129022. PMID 24761231
- [Background] Brimmo FO, Babatunde AO, Ezefuna NN, Kanu MS, Biziyaremye P. The need for more medical schools in medically underserved regions in Africa. Ann Med Surg (Lond). 2022 Nov 17;84:104967. doi: 10.1016/j.amsu.2022.104967. eCollection 2022 Dec. PMID 36426098
- [Background] Pellegrino JL, Charlton N, Goolsby C. "Stop the Bleed" Education Assessment Tool (SBEAT): Development and Validation. Cureus. 2020 Sep 21;12(9):e10567. doi: 10.7759/cureus.10567. PMID 33101813
- [Background] De Buck E, Van Remoortel H, Dieltjens T, Verstraeten H, Clarysse M, Moens O, Vandekerckhove P. Evidence-based educational pathway for the integration of first aid training in school curricula. Resuscitation. 2015 Sep;94:8-22. doi: 10.1016/j.resuscitation.2015.06.008. Epub 2015 Jun 18. PMID 26093230
- [Background] Tse E, Plakitsi K, Voulgaris S, Alexiou GA. Teaching Cardiopulmonary Resuscitation and Defibrillation in Children. Pediatr Emerg Care. 2022 Sep 1;38(9):e1577. doi: 10.1097/PEC.0000000000002815. Epub 2022 Aug 9. No abstract available. PMID 35947075
- [Background] De Buck E, Laermans J, Vanhove AC, Dockx K, Vandekerckhove P, Geduld H. An educational pathway and teaching materials for first aid training of children in sub-Saharan Africa based on the best available evidence. BMC Public Health. 2020 Jun 3;20(1):836. doi: 10.1186/s12889-020-08857-5. PMID 32493323
- [Background] Zideman DA, Singletary EM, Borra V, Cassan P, Cimpoesu CD, De Buck E, Djarv T, Handley AJ, Klaassen B, Meyran D, Oliver E, Poole K. European Resuscitation Council Guidelines 2021: First aid. Resuscitation. 2021 Apr;161:270-290. doi: 10.1016/j.resuscitation.2021.02.013. Epub 2021 Mar 24. PMID 33773828
- [Background] Olmos-Gomez MDC, Ruiz-Garzon F, Pais-Roldan P, Lopez-Cordero R. Teaching First Aid to Prospective Teachers as a Way to Promote Child Healthcare. Healthcare (Basel). 2021 Mar 25;9(4):367. doi: 10.3390/healthcare9040367. PMID 33806034
- [Background] Scerbo MH, Holcomb JB, Taub E, Gates K, Love JD, Wade CE, Cotton BA. The trauma center is too late: Major limb trauma without a pre-hospital tourniquet has increased death from hemorrhagic shock. J Trauma Acute Care Surg. 2017 Dec;83(6):1165-1172. doi: 10.1097/TA.0000000000001666. PMID 29190257
- [Background] Pais-Roldan P, Del Carmen Olmos-Gomez M, Cuevas-Rincon JM, Luque-Suarez M. Study on the Attitudes and Knowledge of Teachers and Future Teachers about Immediate Health Care Measures at School. Eur J Investig Health Psychol Educ. 2022 Jul 20;12(7):854-869. doi: 10.3390/ejihpe12070062. PMID 35877462
- See also: Contains documents for information related to this protocol — https://drive.google.com/drive/folders/1oaz8ewLKW--cX5Nm7Y0I_j0jPhJzwzVS?usp=sharing
- Available data/document: Study Protocol: vanesssatob@gmail.com — https://drive.google.com/drive/folders/1oaz8ewLKW--cX5Nm7Y0I_j0jPhJzwzVS?usp=sharing

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT07110077/Prot_ICF_000.pdf